CLINICAL TRIAL: NCT03457597
Title: A Phase 1, Open-Label, Single-Sequence Crossover Study in Healthy Subjects to Determine the Effect of Relacorilant on Exposure to Probe Substrates for Cytochrome P450s 3A4, 2C8, 2C9, 2C19, and 2D6
Brief Title: Study in Healthy Subjects to Determine the Effect of Relacorilant on Exposure to Probe Substrates for Cytochrome P450s
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CORT125134-126
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-02

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam; Metoprolol; Pioglitazone; Tolbutamide; Omeprazole; relacorilant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Period 1 (Experimental): Period 1 (Study Days 1 to 4): Midazolam hydrochloride and metoprolol tartrate will be given once on Day 1. Pioglitazone hydrochloride, tolbutamide and omeprazole will be given once on Day 2
  Interventions: Drug: Midazolam hydrochloride; Drug: Metoprolol tartrate; Drug: Pioglitazone hydrochloride; Drug: Tolbutamide; Drug: Omeprazole
- Period 2 (Experimental): Period 2 (Study Days 5 to 13): Relacorilant will be given daily from Day 5 to Day 13.
  Interventions: Drug: Relacorilant
- Period 3 (Experimental): Period 3 (Study Days 14 to 17): Midazolam hydrochloride and metoprolol tartrate will be given once on Day 14. Pioglitazone hydrochloride, tolbutamide and omeprazole will be given once on Day 15. Relacorilant will be given daily from Day 14 to Day 17.
  Interventions: Drug: Midazolam hydrochloride; Drug: Metoprolol tartrate; Drug: Pioglitazone hydrochloride; Drug: Tolbutamide; Drug: Omeprazole; Drug: Relacorilant

INTERVENTIONS:
Drug: Midazolam hydrochloride — Midazolam hydrochloride 2.5 mg
  Other Names: Versed
  Arms: Period 1; Period 3
Drug: Metoprolol tartrate — Metoprolol tartrate 100 mg
  Other Names: Lopressor
  Arms: Period 1; Period 3
Drug: Pioglitazone hydrochloride — Pioglitazone hydrochloride 15 mg
  Other Names: Actos
  Arms: Period 1; Period 3
Drug: Tolbutamide — Tolbutamide 500 mg
  Other Names: Orinase
  Arms: Period 1; Period 3
Drug: Omeprazole — Omeprazole 20 mg
  Other Names: Prilosec
  Arms: Period 1; Period 3
Drug: Relacorilant — Relacorilant 350mg
  Other Names: CORT125134
  Arms: Period 2; Period 3

SUMMARY:
This is an open-label, single-sequence, 3-period crossover study conducted in healthy subjects. Eligible subjects will participate in a single treatment period, in which they will receive the following treatments: Day 1, single doses of midazolam and metoprolol; Day 2, single doses of pioglitazone, tolbutamide, and omeprazole; Days 5 to 17, daily doses of relacorilant; Day 14, single doses of midazolam and metoprolol (with relacorilant); and, Day 15, single doses of pioglitazone, tolbutamide, and omeprazole (with relacorilant).

DETAILED DESCRIPTION:
This is an open-label, single-sequence, 3-period crossover study conducted in healthy subjects. Subjects will be screened for eligibility for the study within 21 days before the first dose of study drug based on entrance criteria specified in Section 4. Eligible subjects will participate in a single treatment period, in which they will receive the following treatments:

* Day 1: single doses of midazolam and metoprolol
* Day 2: single doses of pioglitazone, tolbutamide, and omeprazole
* Days 5 to 17: daily doses of relacorilant
* Day 14: single doses of midazolam and metoprolol (with relacorilant)
* Day 15: single doses of pioglitazone, tolbutamide, and omeprazole (with relacorilant) Blood samples will be collected before dosing and at intervals up to 24 hours after each midazolam dose, up to 48 hours after each metoprolol, tolbutamide, and omeprazole dose, and up to 72 hours after each pioglitazone dose for assay of the respective probe substrates and relevant metabolites. Additional samples will be collected during the relacorilant dosing period for assay of relacorilant and metabolites to confirm exposure and at the beginning (before dosing on Day 5) and near the end (Day 14) of the relacorilant dosing period for assay for 4β-OH cholesterol, a biomarker for CYP induction.

Safety and tolerability will be monitored using AEs, clinical laboratory evaluations, 12-lead ECG recordings, vital sign and pulse oximetry measurements, and physical examinations.

Subjects will be admitted to the Clinical Research Unit (CRU) on the morning of Day -1 following an 8-hour fast for baseline assessments and will remain confined until completion of procedures, 72 hours after the last dose of probe substrate and 24 hours after the last dose of relacorilant. Subjects may leave the CRU after safety review on the morning of Day 18. Each subject will have a follow-up (FU) visit 14 ± 2 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the purpose and risks of the study; willing and able to adhere to scheduled visits, treatment plans, laboratory tests, and other study evaluations and procedures.
2. Give written informed consent.
3. Be males or nonpregnant, nonlactating females judged to be in good health, based on the results of medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory findings.
4. Have a body mass index (BMI) between 18 and 32 kg/m2, inclusive, and a body weight more than 50 kg (110 pounds).
5. Be a nonsmoker. Use of nicotine or nicotine-containing products must be discontinued at least 90 days prior to the first dose of study drug.
6. Be willing to comply with study restrictions
7. Have suitable veins for multiple venipuncture/cannulation.
8. Female subjects must be either of nonchildbearing potential (ie, postmenopausal or permanently sterilized) or use highly effective contraception with low user-dependency.

   * The only acceptable method of highly effective contraception with low user-dependency is an intrauterine device (IUD). Use of hormonal contraception (by any route, including intrauterine hormone releasing systems) or hormone replacement therapy is NOT acceptable.

Exclusion Criteria:

1. Be an employee or immediate family member of the Clinical Research Unit or Corcept.
2. Have been previously enrolled in any study of relacorilant.
3. Have multiple drug allergies, or be allergic to any of the components of relacorilant.
4. Have a condition that could be aggravated by glucocorticoid blockade (eg, asthma, any chronic inflammatory condition).
5. Have a history of gastric bypass surgery.
6. Have a history of malabsorption syndrome or previous gastrointestinal surgery, with the exception of appendectomy and cholecystectomy, which could affect drug absorption or metabolism.
7. Current alcohol or substance abuse.
8. In the 2 calendar months before first study drug administration, have donated/lost blood or plasma in excess of 400 mL.
9. In the 30 days before first study drug administration, have participated in another clinical trial of a new chemical entity or a prescription medicine.
10. Have a positive test for alcohol or drugs of abuse at screening or first admission.
11. Have a positive test for exogenous glucocorticoids at screening.
12. Have clinically relevant abnormal findings on vital signs, physical examination, laboratory screening tests, or 12-lead ECG, at screening and/or before first study drug administration, including but not limited to**:

    1. QT interval corrected for heart rate (QTc) using Fridericia's equation (QTcF) >450 ms (from mean of 3 supine ECGs, performed at least 2 minutes apart)
    2. Stage 2 or higher hypertension (supine/semi-recumbent systolic blood pressure [SBP] >160 mmHg, diastolic blood pressure [DBP] >100 mmHg; based on mean of duplicate values recorded at least 2 minutes apart)
    3. Stage 1 hypertension (supine/semi-recumbent SBP 140-160 mmHg, DBP 90-100 mmHg; based on mean of duplicate values recorded at least 2 minutes apart) associated with indication for treatment ie, evidence of end-organ damage, diabetes, or a 10-year cardiovascular risk, estimated using a standard calculator, (eg, QRISK2-2016) greater than 20%
    4. Glomerular filtration rate, estimated using the chronic kidney disease epidemiology (collaboration) (CKD-EPI) method (eGFR; Levey 2009) <60 mL/minute/1.73 m2
    5. Hypokalemia (potassium below lower limit of normal)
    6. Alanine aminotransferase (ALT), aspartate amino transferase (AST), and/or gamma- glutamyltransferase (GGT) >1.5 times the upper limit of normal (ULN)
    7. Seropositive for hepatitis B, hepatitis C, or human immunodeficiency (HIV) viruses **For purposes of qualifying any given subject for study participation, out-of-range values may be repeated once.
13. Have any medical or social reasons for not participating in the study raised by their primary care physician.
14. Have any other condition that might increase the risk to the individual or decrease the chance of obtaining satisfactory data, as assessed by the Investigator.
15. Taken any prohibited prior medication within protocol designated timeframes, such as or including any glucocorticoid, strong inducers, inhibitors or substrates of CYP enzymes involved in drug-drug-interactions, hormonal contraception or hormone replacement therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-28 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve up to the last quantifiable sample (AUC0-tz) | predose to 96 hrs postdose
  Ratio of population geometric means (GMR) for Reference Day (following a single dose with each probe substrate given within a cocktail of probe substrates) and Test Day (following the same dose given to subjects after 10 or 11 days of daily dosing with relacorilant) areas under plasma concentration-time curve up to the last quantifiable sample (AUC0-tz)

SECONDARY OUTCOMES:
Area under plasma concentration-time curve extrapolated to infinity (AUCinf) | predose to 96 hrs postdose
  Ratio of population geometric means (GMR) for Reference Day (following a single dose with each probe substrate given within a cocktail of probe substrates) and Test Day (following the same dose given to subjects after 10 days of daily dosing with relacorilant) areas under plasma concentration-time curve extrapolated to infinity (AUCinf)
Maximum plasma concentration (Cmax) | predose to 96 hrs postdose
  Ratio of population geometric means (GMR) for Reference Day (following a single dose with each probe substrate given within a cocktail of probe substrates) and Test Day (following the same dose given to subjects after 10 days of daily dosing with relacorilant) maximum plasma concentration (Cmax).
Adverse Events | up to 8 weeks
  Safety and tolerability measure by number of subjects who experience adverse events
Safety Labs | up to 8 weeks
  Safety and tolerability measure by number of subjects who experience potential clinically significant changes in safety labs
ECGs | up to 8 weeks
  Safety and tolerability measure by number of subjects who experience potential clinically significant changes in ECGs
Vital Signs | up to 8 weeks
  Safety and tolerability measure by number of subjects who experience potential clinically significant changes in vital signs
Physical Examinations | up to 8 weeks
  Safety and tolerability measure by number of subjects who experience potential clinically significant changes in physical exams

CONTACTS AND LOCATIONS:
Overall Officials: Kirsteen Donaldson, FFPM,DM,FRCP, Study Director — Corcept Therapeutics
Locations (1):
- Celerion, Tempe, Arizona, United States